CLINICAL TRIAL: NCT02541851
Title: Chronic Pain After Surgical Intensive Care Admission: Incidence and Risk Factors: the DOLOCHROREA Study
Acronym: DOLOCHROREA
Status: Terminated | Type: Observational
Why Stopped: Insufficient recruitment leading to selection bias and insufficient data
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Principal Investigator, Guillaume BESCH, M.D., Centre Hospitalier Universitaire de Besancon
Other Study IDs: 15/03
Record Dates: First submitted 2015-09-03; First posted 2015-09-04 (Estimated); Last update posted 2017-08-02 (Actual); Status verified 2017-08

CONDITIONS: Pain, Chronic; Intensive Care, Surgical
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The acute pain remains unfortunately a major health problem in intensive care patients. Several factors, such as cancer, traumatic injuries, surgery, scars, diagnostic or therapeutic procedure, could contribute to an increase in the incidence or in the intensity of acute pain. The acute pain could impact on the prognosis of intensive care patients and on the patients perception of the quality of care.

Moreover, the acute pain could lead to a long-term chronic pain syndrome. The chronic pain after intensive care admission could threaten the physical and psychological recovery after the stay in the intensive care unit (ICU).

If many studies have been conducted to improve the management of the acute pain in the ICU, only few data exist on the incidence and the risk factors of the chronic pain after a stay in a surgical intensive care.

The aim of the DOLOCHROREA study is to assess the incidence and the risk factors of 6-month chronic pain after a stay in our surgical ICU.

ELIGIBILITY:
Inclusion Criteria:

* Admission in the surgical critical care unit of the University Hospital of Besançon from February 2015
* Age over 18 yr old
* Informed consent

Exclusion Criteria:

* Age under 18 yr old
* Death within the first 6 months after the end of the stay in the surgical intensive unit of the University Hospital of Besançon
* Glasgow Coma Score under 8 at admission and/or at discharge
* Planned admission after elective surgery
* Medical history of cognitive disorder
* Refuse to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted in the surgical critical care unit of the Centre Hospitalier Universitaire de Besançon, France.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Incidence of chronic pain | 6 months
  Pain is defined by The International Association for the Study of Pain (IASP) as "an unpleasant sensory and emotional experience associated with actual or potential tissue damage". Pain exceeding the average period of healing of 2 to 3 months and ceasing to serve any apparent protective function is defined as chronic pain. The incidence of chronic pain will be assessed by using a validated french version of the Brief Pain Inventory during a phone call at 6 month after the end of the stay in our intensive care unit.

SECONDARY OUTCOMES:
Incidence of anxiety and depression | 6 months
  The incidence of anxiety and depression at 6 months after the end of the stay in our intensive care unit will be assessed by using a validated french version of the Hospital Anxiety and Depression (HAD) scale during a phone call.
Incidence of neuropathic pain | 6 months
  The incidence of neuropathic pain at 6 months after the end of the stay in our intensive care unit will assessed by using the DN4 tool during a phone call.

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume Besch, M.D., Principal Investigator — Centre Hospitalier Universitaire de Besançon
Locations (1):
- Centre Hospitalier Universitaire de Besançon, Besançon, France

REFERENCES:
- [Background] Battle CE, Lovett S, Hutchings H. Chronic pain in survivors of critical illness: a retrospective analysis of incidence and risk factors. Crit Care. 2013 May 29;17(3):R101. doi: 10.1186/cc12746. PMID 23718685